CLINICAL TRIAL: NCT04943809
Title: Comparison of Visual Outcomes After Implantation of the POD 26P AY FT (PhysIOL) and the POD 26P AY F (PhysIOL)
Brief Title: Comparison of Visual Outcomes After Implantation of the POD FT and the POD F
Acronym: PoyPODF/FT
Status: Completed | Type: Observational
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Poyales/POD FT - POD F
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Cataract
Keywords: Hydrophilic; Toric; intraocular lens; cataract; trifocal; BVI Medical
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD 26P AY FT: 26 patients with corneal astigmatism higher than 1.0D in both eyes and lower than 2.5D and will be implanted with the POD 26P AY FT
  Interventions: Device: POD 26P AY FT
- POD 26P AY F: 26 patients with corneal astigmatism lower than 1.0D in both eyes will be implanted with the POD 26P AY F
  Interventions: Device: POD 26P AY F

INTERVENTIONS:
Device: POD 26P AY FT — Routine cataract surgery
  Groups: POD 26P AY FT
Device: POD 26P AY F — Routine cataract surgery
  Groups: POD 26P AY F

SUMMARY:
There is no difference of the photic phenomena in the two groups.

The study will be a prospective non-randomised controlled study. The target is then to determine the equivalence in the glare. Assumption of Type I error is p=0.05 as level of significance and Type II error is alpha=0.8 as power.

DETAILED DESCRIPTION:
The study will be a prospective non-randomised controlled study. The target is then to determine the equivalence in the glare. Assumption of Type I error is p=0.05 as level of significance and Type II error is alpha=0.8 as power.

We used the 'TrialSize' package of the R software. Here are the parameters defined for the sample size calculation:

1. Alpha: 0.05
2. Power : 0.90
3. Two sided test
4. Equal group allocation
5. Standard deviation for the two groups (POD 26P AY F et POD 26P AY FT) equal to 0.10
6. Expected mean for the two groups (POD 26P AY F et POD 26P AY FT) equal to 0.89 (true difference between the means equal 0)
7. An equivalence limit of 0.05, 0.10 and 0.15 Equivalence limit: 0.15 In order to show no difference between these two groups, 12 patients by groups are needed. With a drop-out of 15%, we obtain 30 patients (15 patients by group) to recruit in order to obtain 24 valuable patients.

Equivalence limit: 0.10 In order to show no difference between these two groups, 26 patients by groups are needed. With a drop-out of 15%, we obtain 62 patients (31 patients by group) to recruit in order to obtain 52 valuable patients.

This total number of subjects with such requirement is 26 patients in each group.

Group 1 will be made of 26 patients with corneal astigmatism higher than 1.0D in both eyes and lower than 2.5D and will be implanted with the POD 26P AY FT and Group 2 will be made of 26 patients with corneal astigmatism lower than 1.0D in both eyes.

Interim analysis after the 12th patient of each group will have completed the last follow-up will be achieved to confirm the equivalence with the equivalence limit of 0.15.

The POD platform in 26 % (non toric version) is available since 2008 in the monofocal version and since 2012 in the toric one (POD 6P AY T, Ankoris®, PhysIOL).The so-called POD design is characterised by two symmetrical bifid haptics with opened loops that provide four points of support to ensure IOL stability in the capsular bag. The dual C-loop profile shortens the loops, thus improving the pliability of the implant during its injection through a micro-incision. These shortened loops should permit a clockwise or anticlockwise rotary motion and should facilitate the comfortable fitting of the implant orientation after unfolding without elastic-restoring torque. The double C-loop POD design offers 4 support points for the implant within the capsule and ensures its stability. The V-shape of the upper and lower haptics together with the flexibility of the implant allow the loop separation angle to be adjusted and ensure the most accurate adaptation to the capsular bag size. A finite element structural analysis of the implant showed that the elasticity at the distal part of the loop prevents the constraints from being transmitted onto the optical portion of the implant. The trifocal optic is associated to the POD platform and is made of 26 % raw material.

The rotational stability of this non toric version has been clinically investigated on 117 consecutive eyes 1 week, 3 weeks, 3 and 12 months after implantation. The absolute rotation of the lens averaged 2.5 ± 2.6°. The position of the center of the implant relative to the pupillary center expressed by a vector was 0.01 mm at 70°.

The investigational product (POD 26P AY FT) is CE labeled since January 2014. Main IOL features are:

* Biconvex toric aspheric (-0.11um SA) blue-blocking, hydrophilic acrylic IOL with 26% equlibrium water content, implantable through ≥ 2.2mm incision.
* 4-point haptic design
* 6 mm of optical diameter / 11.4 mm of total diameter
* Dioptric range (SE): 6 to 35 D by 0.5 D increments
* Cylinders at the IOL plane: 1, 1.5, 2.25, 3, 3.75, 4.5, 5.25, 6 D
* Addition +1.75D / +3.5 D

The control product (POD 26P AY F) is CE labeled since 2010. Main IOL features are:

* Biconvex, aspheric (-0.11um SA) blue-blocking, hydrophilic acrylic IOL with 26% equlibrium water content, implantable through ≥ 2.2mm incision.
* 4-point haptics design which minimizes decentration and optimizes the rotational stability
* 6 mm of optical diameter / 11.4 mm of total diameter
* Dioptric range (SE): 6 to 35 D by 0.5 D increments
* Addition +1.75D / +3.5 D

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Preoperative Corneal astigmatism < 0.75 D
* Age 21 and older
* Visual Acuity > 0.05
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.
* Patient willing multifocal implantation and with realistic expectations.

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome, floppy iris syndrome, corneal pathologies, retinal pathology (diabetic maculopathy, myopic maculopathy, age related macular degeneration...)
* Previous ocular surgery or trauma.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients undergoing routine cataract surgery. The study participants receive a bilateral implantation of trifocal intraocular lenses. Depending on the preoperative corneal astigmatism, the patients receive either non-toric trifocal IOLs (POD F) or toric trifocal IOLs (POD FT) in both eyes.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Determine the equivalence of the glare | 3 Months
  The primary endpoint is to show statistically equivalent outcomes on glare at the 3 months follow up visit. A significance level of p = 0.05 will be considered statistically significant.

SECONDARY OUTCOMES:
Measurement of far, intermediate and near visual acuity | 6 Months
  The secondary objective is to measure far, intermediate and near visual acuity of the POD AY 26P FT with respect to the POD AY 26P F.
Refraction | 6 Months
  The secondary objective is to measure the refraction of the POD AY 26P FT with respect to the POD AY 26P F.
Centration | 6 Months
  The secondary objective is to measure the centration of the POD AY 26P FT with respect to the POD AY 26P F.
Rotational stability | 6 Months
  The secondary objective is to measure the rotational stability of the POD AY 26P FT with respect to the POD AY 26P F.
Equivalence of the visual acuity and the contrast sensitivity | 6 Months
  The secondary objective is to determine the equivalence of the visual acuity of the POD AY 26P FT with respect to the POD AY 26P F.
Equivalence of the visual acuity and the contrast sensitivity | 6 Months
  The secondary objective is to determine the contrast sensitivity at far of the POD AY 26P FT with respect to the POD AY 26P F.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Poyales Galan, PhD, Principal Investigator — CEIC Hospital Clinical San Carlos
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chassain C, Pagnoulle C, Gobin L, Rozema J. [Evaluation of a new intraocular lens platform: centration and rotational stability]. J Fr Ophtalmol. 2013 Apr;36(4):336-42. doi: 10.1016/j.jfo.2012.04.012. Epub 2013 Jan 24. French. PMID 23352708
- [Result] Visser N, Bauer NJ, Nuijts RM. Toric intraocular lenses: historical overview, patient selection, IOL calculation, surgical techniques, clinical outcomes, and complications. J Cataract Refract Surg. 2013 Apr;39(4):624-37. doi: 10.1016/j.jcrs.2013.02.020. PMID 23522584
- [Result] de Vries NE, Nuijts RM. Multifocal intraocular lenses in cataract surgery: literature review of benefits and side effects. J Cataract Refract Surg. 2013 Feb;39(2):268-78. doi: 10.1016/j.jcrs.2012.12.002. PMID 23332253
- [Result] Wolffsohn JS, Jinabhai AN, Kingsnorth A, Sheppard AL, Naroo SA, Shah S, Buckhurst P, Hall LA, Young G. Exploring the optimum step size for defocus curves. J Cataract Refract Surg. 2013 Jun;39(6):873-80. doi: 10.1016/j.jcrs.2013.01.031. PMID 23688874
- [Result] Sheppard AL, Shah S, Bhatt U, Bhogal G, Wolffsohn JS. Visual outcomes and subjective experience after bilateral implantation of a new diffractive trifocal intraocular lens. J Cataract Refract Surg. 2013 Mar;39(3):343-9. doi: 10.1016/j.jcrs.2012.09.017. Epub 2013 Jan 16. PMID 23332118
- [Result] Cochener B, Vryghem J, Rozot P, Lesieur G, Heireman S, Blanckaert JA, Van Acker E, Ghekiere S. Visual and refractive outcomes after implantation of a fully diffractive trifocal lens. Clin Ophthalmol. 2012;6:1421-7. doi: 10.2147/OPTH.S32343. Epub 2012 Sep 3. PMID 22969289
- [Result] Roensch MA, Charton JW, Blomquist PH, Aggarwal NK, McCulley JP. Resident experience with toric and multifocal intraocular lenses in a public county hospital system. J Cataract Refract Surg. 2012 May;38(5):793-8. doi: 10.1016/j.jcrs.2011.11.043. Epub 2012 Mar 15. PMID 22425363
- [Result] Visser N, Nuijts RM, de Vries NE, Bauer NJ. Visual outcomes and patient satisfaction after cataract surgery with toric multifocal intraocular lens implantation. J Cataract Refract Surg. 2011 Nov;37(11):2034-42. doi: 10.1016/j.jcrs.2011.05.041. Epub 2011 Sep 22. PMID 21940140
- [Result] Bellucci R, Bauer NJ, Daya SM, Visser N, Santin G, Cargnoni M, Nuijts RM; Lisa Toric Study Group. Visual acuity and refraction with a diffractive multifocal toric intraocular lens. J Cataract Refract Surg. 2013 Oct;39(10):1507-18. doi: 10.1016/j.jcrs.2013.04.036. PMID 24075158
- [Result] Alfonso JF, Knorz M, Fernandez-Vega L, Rincon JL, Suarez E, Titke C, Kohnen T. Clinical outcomes after bilateral implantation of an apodized +3.0 D toric diffractive multifocal intraocular lens. J Cataract Refract Surg. 2014 Jan;40(1):51-9. doi: 10.1016/j.jcrs.2013.06.026. PMID 24355720
- [Result] Ferreira TB, Marques EF, Rodrigues A, Montes-Mico R. Visual and optical outcomes of a diffractive multifocal toric intraocular lens. J Cataract Refract Surg. 2013 Jul;39(7):1029-35. doi: 10.1016/j.jcrs.2013.02.037. Epub 2013 May 13. PMID 23680631
- [Result] Knorz MC, Rincon JL, Suarez E, Alfonso JF, Fernandez-Vega L, Titke C, Kohnen T, Tucker S. Subjective outcomes after bilateral implantation of an apodized diffractive +3.0 D multifocal toric IOL in a prospective clinical study. J Refract Surg. 2013 Nov;29(11):762-7. doi: 10.3928/1081597X-20131021-06. PMID 24203808